CLINICAL TRIAL: NCT05392335
Title: Effects Of Myofascial Stretch With And Without Functional Massage On Spasticity And Gross Motor Function In Children With Cerebral Palsy
Brief Title: Myofascial Stretch With And Without Functional Massage In Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0705
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy, Functional Massage, Myofacial Stretch
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myofascial stretch group (Active Comparator): Patients will be given myofascial stretch
  Interventions: Other: Myofascial stretch
- Functional massage along with myofascial stretch group (Experimental): patients will be given functional massage along with myofascial stretching
  Interventions: Other: Myofascial stretch; Other: Functional massage along with myofacial stretch

INTERVENTIONS:
Other: Myofascial stretch — Myofascial stretch will be applied at hip adductors, hamstrings and calf muscles for 10 -15 repetitions on each muscle. 2-3 sessions will be performed in a week for 8 weeks.
Other: Functional massage along with myofacial stretch — In this group during the first 20 minutes, ten minutes FM will be applied to each lower extremity of the subject. The muscle groups to which FM would be applied were hip adductors, hamstrings and calf muscles. During the remaining period traditional physiotherapy involving myofascial strecth will be given. 2-3 session will be performed in a week for 8 weeks.
  Arms: Functional massage along with myofascial stretch group

SUMMARY:
Cerebral palsy is one of the most common childhood disabilities, and it occurs with an incidence of 2-2.5 per 1000 living births. Children with CP have various impairments including neuromuscular and musculoskeletal problems such as spasticity, dyscoordination, loss of selective motor control, and weakness. CP can be classified according to the severity of motor deficits as mild, moderate, or severe. Several other classification systems exist based on the pathophysiology, etiology, and distribution of motor deficits. The aim of the study to evaluate the effects of functional massage and myofascial stretch on spasticity and motor function of CP Children. Study will be conducted in 22 patients in experimental and control group. Pre and Post values will be evaluated. The tools used will be Modified Ashworth Scale (MAS) and Gross Motor Function Measure (GMFM). The significance of this study is that it will define for us that to how much extent we can improve the Spastic and painful condition of lower limb of CP child. Data will be analyzed using SPSS 22.0 mean and standard deviation will be calculated. Appropriate the statistical test will be used after checking normality of data.

ELIGIBILITY:
Inclusion Criteria:

* Age of 6 and 12 year
* Both genders
* Children between level Ⅰ- Ⅳ based on Gross Motor Classification System(GMFCS)

Exclusion Criteria:

* The existence of dyskinesia or dystonia
* History of muscle lengthening surgery
* Presence of uncontrolled seizures

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change in scores of Modified Ashworth scale | Baseline and 8th week
  The modified Ashworth scale(MAS) is a 6-point rating scale that is used to measure muscle tone.(20) The reliability of the modified Ashworth scale was very good (κw = .84 for inter rater and .83 for intra-rater comparisons)
Change in scores of GMFM 88 | Baseline and 8th week
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline. However, most of the items have specific descriptors for each score. It is imperative that the guidelines contained in the manual be used for scoring each item. SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes 9 (or leave blank) = not tested (NT)

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmood Q, Habibullah S, Babur MN. Potential effects of traditional massage on spasticity and gross motor function in children with spastic cerebral palsy: A randomized controlled trial. Pak J Med Sci. 2019 Sep-Oct;35(5):1210-1215. doi: 10.12669/pjms.35.5.478. PMID 31488980
- [Background] BİNGÖL H, YILMAZ Ö. Effects of functional massage on spasticity and motor functions in children with cerebral palsy: a randomized controlled study. Journal of Exercise Therapy and Rehabilitation. 2018;5(3):135-42.
- [Background] Bingöl H, Akaras E, Kocaman H. The effects of massage therapy on symptoms related cerebral palsy in children with cerebral palsy: A systematic review. Journal of Clinical Medicine of Kazakhstan. 2020;4(58):6-14.
- [Background] Kuruma H, Takei H, Nitta O, Furukawa Y, Shida N, Kamio H, et al. Effects of Myofascial Release and Stretching Technique on Range of Motion and Reaction Time. Journal of Physical Therapy Science. 2013;25(2):169-71.